CLINICAL TRIAL: NCT04493294
Title: Low Dose Whole Lung Radiotherapy for Older Patients With Coronavirus 19 Disease (COVID-19) Pneumonitis: Practical Protocol by the International Geriatric Radiotherapy Group
Brief Title: Low Dose Whole Lung Radiotherapy for Older Patients With COVID-19 Pneumonitis
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: International Geriatric Radiotherapy Group (Other)
Collaborators: Brigitta G. Baumert (Unknown)
Responsible Party: Principal Investigator, Nam Nguyen, President, International Geriatric Radiotherapy Group
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IGRG01
Record Dates: First submitted 2020-07-29; First posted 2020-07-30 (Actual); Last update posted 2020-07-30 (Actual); Status verified 2020-07

CONDITIONS: COVID-19 Pneumonitis
Keywords: COVID-19; pneumonitis; whole lung radiotherapy; low dose
MeSH Terms: conditions — COVID-19; Pneumonia

STUDY DESIGN:
Intervention Model Description: Using low dose whole lung radiotherapy to older patients who develop COVID-19 pneumonitis to improve their survival compared to historical data
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Radiation: Low dose whole lung radiotherapy for older patients with COVID-19 pneumonitis — Low dose whole lung radiotherapy may decrease the cytokines storm related to the viral infection and may improve survival by decreasing the need for artificial ventilation

SUMMARY:
Low dose whole lung radiotherapy may improve survival of older patients with COVID-19 pneumonitis

DETAILED DESCRIPTION:
Background: Coronavirus disease 19 (COVID-19) carry a high mortality rate among older patients and minorities such as ethnic Africans and Latinos. The chronic baseline systemic inflammation of older patients and minorities may make them more vulnerable to the cytokines storm generated by the viral infection in addition to preexisting co-morbidity.

Even though multiple organs failure result from the cytokine storm, pneumonia and respiratory failure often lead to death. Low dose whole lung radiotherapy (LDWLRT) may modulate the inflammatory response and may decrease the need for artificial ventilation, thus improving mortality rate.

Methods: A phase I-II prospective trials enrolling 500 patients, 65 years old or older from 26 countries will be conducted to investigate the impact of LDWLRT on mortality rate of COVID-19 patients. The patients who will be selected would have developed pneumonias but did not require artificial ventilation. These patients will be followed for a year after receiving this treatment. Their physical activities will be monitored through the ordinal scale and will be correlated with their cytokines status and oxygen saturation rate to assess the impact of the residual inflammation on their daily life. Mortality rates between different ethnic group will be compared and correlated with their cytokines response to the virus and number of co-morbidities.

Discussion and importance of the study: We postulate that LDWLRT may improve survival rates of all patients by preventing the need for artificial ventilation which is associated with a high mortality. The inflammatory response between different ethnic groups before and following radiotherapy will be valuable to serve as baseline for future prospective pandemic studies as it has not been reported before.

ELIGIBILITY:
Inclusion Criteria:

* 65 years-old or older patients with proven COVID-19 pneumonitis who may or may not require oxygen

Exclusion Criteria:

* Patients with pneumonia who do not have a diagnosis of COVID-19 infection, patients with COVID-19 pneumonitis who require artificial ventilation or hemodynamically unstable to undergo radiotherapy or consent cannot be obtained either through the patient or power of attorney or patients already enrolled in another clinical trial

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2020-11 (Estimated); Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Mortality rate | One year
  Comparing mortality rate of the whole group of patients treated with low dose whole lung radiotherapy with historical data

SECONDARY OUTCOMES:
Mortality rate | One year
  Comparison mortality rate of different ethnic groups treated with whole lung radiotherapy for COVID-19 pneumonia
Duration of hospitalization | One year
  Duration of hospitalization for the whole group and different groups with or without oxygen requirement
Time to recovery | One month
  Ordinal scale at the time of radiotherapy and 28 days later
Oxygen saturation rate | One year
  Correlation between oxygen saturation rate and ordinal scale at different times following radiotherapy
Patient inflammatory status | One year
  Biomarkers for inflammation such as Interleukin 6 will be monitored and correlated with ordinal scale at different times following radiotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Brigitta G Baumert, M.D.Ph.D, Principal Investigator — Institute of Radiation Oncology, Cantonal hospital Graubuenden, Chur, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided
There are over 40 people involved in the study, we need their approval before data sharing

REFERENCES:
- [Background] Lara PC, Burgos J, Macias D. Low dose lung radiotherapy for COVID-19 pneumonia. The rationale for a cost-effective anti-inflammatory treatment. Clin Transl Radiat Oncol. 2020 Apr 25;23:27-29. doi: 10.1016/j.ctro.2020.04.006. eCollection 2020 Jul. PMID 32373721
- [Background] Lara PC, Nguyen NP, Macias-Verde D, Burgos-Burgos J, Arenas M, Zamagni A, Vinh-Hung V, Baumert BG, Motta M, Myint AS, Bonet M, Popescu T, Vuong T, Appalanaido GK, Trigo L, Karlsson U, Thariat J. Whole-lung Low Dose Irradiation for SARS-Cov2 Induced Pneumonia in the Geriatric Population: An Old Effective Treatment for a New Disease? Recommendation of the International Geriatric Radiotherapy Group. Aging Dis. 2020 May 9;11(3):489-493. doi: 10.14336/AD.2020.0506. eCollection 2020 May. PMID 32489696